CLINICAL TRIAL: NCT06341075
Title: Real-World Study of Magnetic Resonance-guided Laser Interstitial Thermal Therapy for Patients With Drug-resistant Epilepsy
Brief Title: Real-World Study of Magnetic Resonance-guided Laser Interstitial Thermal Therapy for Drug-resistant Epilepsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2024-053-02
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Drug Resistant Epilepsy
Keywords: MRgLITT; Drug-resistant Epilepsy; Seizure Control; Functional Preservation; Real-world STUDY
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic Resonance-guided Laser Interstitial Thermal Therapy (MRgLITT) (Experimental): Novel, minimally invasive MRgLITT.
  Interventions: Device: Magnetic Resonance-guided Laser Interstitial Thermal Therapy (MRgLITT)
- Open Surgery (OS) (No Intervention): Traditional OS, including ATL, SAH and so on.

INTERVENTIONS:
Device: Magnetic Resonance-guided Laser Interstitial Thermal Therapy (MRgLITT) — MRgLITT employs laser energy delivered through a stereotactically placed laser applicator to precisely ablate the epileptogenic tissue.
  Arms: Magnetic Resonance-guided Laser Interstitial Thermal Therapy (MRgLITT)

SUMMARY:
The goal of the real-world study is to evaluate the long-term seizure control outcomes, postoperative complications, long term impact on cognitive, memory function outcomes, quality-of-life measures, and healthcare resource utilization of magnetic resonance-guided laser interstitial thermal therapy (MRgLITT) on patients with drug-resistant epilepsy (DRE).

DETAILED DESCRIPTION:
Epilepsy, a complex neurological disorder characterized by recurrent seizures, affects millions of individuals worldwide, challenging both patients and healthcare providers. The main indication for the epilepsy surgery is the drug resistance as per the consensus from the Task Force of the International League Against Epilepsy (ILAE). Traditional open surgery is an established treatment for drug-resistant epilepsy (DRE), but has limitations such as invasiveness and long recovery times. With the significant advancements of technology, the minimally invasive therapeutic approaches have emerged, among which Magnetic Resonance-guided Laser Interstitial Thermal Therapy (MRgLITT) stands out as a promising intervention. It provides targeted ablation of epileptogenic tissue while preserving healthy brain regions. Understanding MRgLITT's comprehensive value for DRE is of increasing interest.

This real-world study aims to comprehensively evaluate the clinical outcomes, safety profiles, and cost-effectiveness of MRgLITT in patients with DRE. The results of this clinical trial protocol are expected to serve as a comprehensive guide for researchers, clinicians, and stakeholders interested in the treatment of DRE using MRgLITT. We believe this study can influence future treatment strategies, leading to improved outcomes and enhanced quality of life for individuals with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 75 (provided that rigorous prior studies have been done to suggest appropriate dosing for ages 12 and above);
* Patients or the assents are able to provide informed consent;
* Ability to keep accurate seizure diaries;
* Complete presurgical evaluation information;
* Meets the 2009 ILAE definition of DRE (Failure of adequate trials of two tolerated and appropriately chosen and used AED schedules (whether as monotherapy or in combination) to achieve sustained seizure freedom) ;

Exclusion Criteria:

* Subjects with significant progressive disorders or unstable medical conditions requiring acute intervention;
* Clinically relevant abnormalities in bloodwork detected (e.g., rising or new onset 3X liver function tests [LFTs]);
* Active suicidal plan/intent in the past 6 months, or a history of suicide attempt in the last 2 years, or more than 1 lifetime suicide attempt;
* A psychiatric disorder where changes in pharmacotherapy are needed or anticipated during the study;
* Diagnosed with intracranial space-occupying lesions or dual pathology by neuroimaging inspection;
* Women who are pregnant, planning to become pregnant during the study period, or currently breastfeeding may be excluded due to the potential risks associated with surgery and anesthesia;
* Patients with a history of previous brain surgery, including prior epilepsy surgery, that may interfere with the study objectives or confound the interpretation of results may be excluded;
* Any condition that may impact a patient's ability to follow study procedures or patient's safety, based on what is known about the pharmacology/toxicology profile of the trial agent(s);

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Seizure-freedom rate | 6-month, 1-year and 2-year after surgery
  Percentage

SECONDARY OUTCOMES:
Seizure frequency reduction | 6-month, 1-year and 2-year after surgery
  Times/Months
ILAE classification of outcome | 6-month, 1-year and 2-year after surgery
  International League Against Epilepsy (ILAE) Outcome Scale. The scale ranges from 1 to 6. The higher value indicates more frequency seizures.
Seizure severity | 6-month, 1-year and 2-year after surgery
  National Hospital Seizure Severity Scale (NHS3). The scale generates a score from 1 to 27. Higher score indicates more severer seizures.
Rate of mild complications | Within 1 month after surgery
  Percentage
Cognitive function evaluation | 6-month, 1-year and 2-year after surgery
  Multiple Ability Self-Report Questionnaire (MASQ). The questionnaire ranges from 38 to 190. Higher score indicates more severer cognitive dysfunction.
Memory function evaluation | 6-month, 1-year and 2-year after surgery
  Memory Functioning Scale Self-Report (MFS-S). The questionnaire ranges from 0 to 42. Higher score indicates more severer memory dysfunction.
The quality of life | 6-month, 1-year and 2-year after surgery
  The EuroQol 5 Dimension 5 Level (ED-5Q-5L). The questionnaire ranges from 0 to 100. Higher score indicates better quality of life.
Length of hospital stay | Within 1 month after surgery
  Days
Rate of reoperations | 6-month, 1-year and 2-year after surgery
  Percentage
Rate of antiepileptic drug reduction or withdrawn | 6-month, 1-year and 2-year after surgery
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zhang, Dr., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact jiajiemo@foxmail.com

REFERENCES:
- [Result] Mo J, Guo Z, Wang X, Zhang J, Hu W, Shao X, Sang L, Zheng Z, Zhang C, Zhang K. Magnetic resonance-guided laser interstitial thermal therapy vs. open surgery for drug-resistant mesial temporal lobe epilepsy: a propensity score matched retrospective cohort study. Int J Surg. 2024 Jan 1;110(1):306-314. doi: 10.1097/JS9.0000000000000811. PMID 37800596